CLINICAL TRIAL: NCT02980549
Title: Determining the Incidence of Parasomnias (PS) and Emergence Delirium (ED)in the American Family Children's Hospital Patient Population
Brief Title: How Common Are Sleep Disorders and Problems With Emergence From Anesthesia in Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0116
Record Dates: First submitted 2015-05-05; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Emergence Delirium; Parasomnias
MeSH Terms: conditions — Emergence Delirium; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: children's sleep habits questionnaire — survey of children's sleep habits completed by parent

SUMMARY:
Emergence delirium (ED), also called emergence agitation or post-anesthetic excitement, is defined as a dissociated state of consciousness, occurring on awakening from general anesthesia, in which children exhibit psychomotor agitation, crying and thrashing and are not consolable for a period of time, usually 5-15 minutes. Emergence delirium is a common problem in pre-school children, with estimates of the incidence ranging from 10-70% of children in this age group. These children are agitated, seemingly unaware of their surroundings, and typically do not respond to parents or caregivers. They are therefore at risk for self-inflicted traumatic injury and complications secondary to disruptions of intravenous lines, surgical incisions, or drains. Children with ED typically require more resources in the postoperative period than children who do not exhibit ED. Predicting the likelihood of ED would allow for better allocation of resources in the post-anesthetic care unit (PACU).

The peak incidence of ED in children occurs in the same age range at which the peak incidence of parasomnias (PS) occurs. The description of parasomnias is strikingly similar to the description of ED; the American Academy of Sleep Medicine defines parasomnias as "undesirable physical events or experiences that occur during entry into sleep, within sleep or during arousals from sleep." Parasomnias can be diagnosed using a sleep questionnaire.

The purpose of this pilot study is to determine the incidence of ED and PS in our population, in order to determine the number of patients necessary to enroll in a larger study to either confirm or reject the hypothesis that ED and PS are correlated.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients age 1-6 (inclusive) scheduled for elective ENT or urologic surgery
2. ASA I or II
3. Presence of a caregiver who is familiar with the child's sleep history

Exclusion Criteria:

1. Autism
2. Severe developmental delay
3. Children receiving clonidine
4. Medication for seizures
5. Children who have received ED treatment prior to a diagnosis of ED (clonidine, dexmedetomidine, or propofol)

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One hundred children age 1-6, ASA PS I or II, undergoing surgery by either elective otolaryngology (ENT) (including but not limited to: tonsillectomy, adenoidectomy, and lymph node biopsy) or elective urologic surgery (including but not limited to: circumcision, cystoscopy and related procedures, orchidopexy or hernia), requiring intravenous line placement, at American Family children's Hospital at the University of Wisconsin will be enrolled in the study. The child's caregiver will complete a sleep questionnaire prior to anesthesia and surgery. From the time the anesthetic is discontinued, after surgery, a study coordinator will observe the child's emergence from anesthesia and rate emergence using the PAED scale every 5 minutes until the child is awake.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of parasomnias (PS) and emergence delirium (ED) in children | 6 months

SECONDARY OUTCOMES:
score on Childrens Sleep Habits Questionnaire correlated with ED | 6 months

IPD SHARING:
Plan to Share IPD: No